CLINICAL TRIAL: NCT01381289
Title: VX-770 Expanded Access Program (EAP)
Brief Title: VX-770 Expanded Access Program
Status: Approved for marketing | Type: Expanded Access
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX11-770-901
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

INTERVENTIONS:
Drug: VX-770 — 150 mg tablet, oral use, twice daily every 12 hours (q12h)

SUMMARY:
The purpose of this expanded access program is to provide VX-770 prior to its commercial availability to people with cystic fibrosis (CF) who have at least one copy of the G551D-CFTR mutation and who are in critical medical need and who are not eligible for participation in other Vertex-sponsored studies.

DETAILED DESCRIPTION:
VX-770, a compound being developed by Vertex Pharmaceuticals Incorporated (Vertex) for the treatment of CF, is an orally bioavailable small molecule that targets the underlying defect in CF, the dysfunctional CFTR protein. In Phase 3 studies of VX-770 in patients with CF and a G551D CFTR mutation, improvements in CFTR function (measured by reduction in sweat chloride concentration) and improvements in lung function were observed.

Patients who are interested in the VX-770 Expanded Access should contact their CF physician about participation.

Physicians interested in participating as a site should contact 800-745-4484.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF, with a sweat chloride >60 mmol/L OR 2 CF-causing mutations AND chronic sinopulmonary disease OR gastrointestinal/nutritional abnormalities.
* Have the G551D-CFTR mutation in at least 1 allele
* Will be aged 6 years or older on the date of signed informed consent form
* Highest FEV1 in the 6 months prior to screening is ≤ 40% predicted value or patient is documented to be active on the lung transplant wait list

Exclusion Criteria:

* If female, currently pregnant
* Abnormal liver function, at screening on recent clinical laboratory testing, defined as >3 × upper limit of normal (ULN), of any 3 or more of the following: AST, ALT, GGT, serum alkaline phosphatase, total bilirubin
* Is currently requiring invasive mechanical ventilation
* Is currently participating, or has participated in the past 30 days in another therapeutic or clinical study

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult